CLINICAL TRIAL: NCT01720069
Title: A Randomised Double-blind, Parallel Group, Dose-ranging Study to Evaluate the Efficacy and Safety of VR506 From a New Dry Powder Inhaler in Subjects With Severe Persistent Asthma Requiring Oral Corticosteroid Therapy.
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of VR506 Using a New Inhaler for the Treatment of Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vectura Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VR506/2/004
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Dose 1 VR506 (Active Comparator): VR506 inhalation powder delivered via a new dry powder inhaler device
  Interventions: Drug: VR506
- Dose 2 VR506 (Active Comparator): VR506 inhalation powder delivered via a new dry powder inhaler device
  Interventions: Drug: VR506
- Dose 3 VR506 (Active Comparator): VR506 inhalation powder delivered via a new dry powder inhaler device
  Interventions: Drug: VR506

INTERVENTIONS:
Drug: VR506 — VR506 inhalation powder delivered via a new dry powder inhaler device

SUMMARY:
To evaluate the clinical efficacy, safety, tolerability and dose-response relationship, using oral corticosteroid (OCS) modulation, of 3 different doses of VR506 using a twice daily regimen from a new dry powder inhaler (nDPI) for 16 weeks in subjects with severe persistent asthma requiring OCS therapy, i.e. Step 5 treatment as defined by modified Global Initiative for Asthma (GINA) guidelines 2011.

ELIGIBILITY:
Inclusion:

* Written informed consent
* Adolescents aged 12-17 years & adults aged 18-65 years (both inclusive)
* Documented clinical history of severe asthma requiring prednisone/prednisolone therapy, high-intensity treatment ICS, OCS, LABA
* Stable OCS dose for ≥7 days before Screening Visit & during Screening Period.
* At least 80% compliant w/regular asthma medication per investigator at end of Screening Period
* Documented asthma reversibility within 5 yrs prior to/during Screening Period, or diagnosis of asthma that is incontrovertible per investigator
* Ability to use nDPI correctly, per investigator's review of completed inhaler operation checklist
* Ability to use eDiary correctly, assessed by investigator at end of Screening Period
* Ability to comply w/study procedures, including blood sampling
* Ability to perform technically satisfactory pulmonary function tests
* Available to complete all study visits before 12 noon
* BMI of 16-26 kg/m2 in adolescents and 18-32 kg/m2 in adults
* Oral PIF ≥40 L/min, using an appropriate device set to match resistance of inhaler
* Good health, except for presence of asthma, per medical history/physical examination
* Negative drug/alcohol/urine cotinine screen. Subjects must test negative for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, cotinine, ethanol & opiates (unless given as prescription medicine)
* Non-smokers or ex-smokers with a smoking history of less than 10 pack-yrs (e.g. <20 cigarettes per day for 10 years or <40 cigarettes per day for 5 years) & stopped smoking for at least 1 year prior to Screening Visit. Smoking will not be permitted throughout study
* Female subjects of child-bearing potential must be using medically acceptable forms of contraception [abstinence, hormonal (oral/implant/transdermal/injection), in use for ≥3 consecutive months before first dose of study medication, double barrier (condom w/spermicide, or diaphragm w/spermicide), IUD, or vasectomised partner (≥6 months since vasectomy)].

Exclusion:

* Regular use (≥3 times/wk) of topical steroids to treat dermatitis/rhinitis/allergic conjunctivitis, within 28 days of Screening Visit
* Subjects who have/who have had, an upper/lower respiratory tract infection within 28 days of Screening Visit
* Subjects w/"brittle asthma
* Subjects w/asthma that required admission to an ICU and/or ventilation within previous 12 months
* Subjects whose comorbidities, per investigator's opinion, are major contributors to their respiratory symptoms (e.g. COPD, bronchiectasis, dysfunctional breathlessness, vocal cord dysfunction, gastro-oesophageal reflux)
* Previously/currently diagnosed as having Churg-Strauss syndrome
* Previously/currently diagnosed as having pulmonary eosinophilia
* History of lung cancer
* Subjects w/current diagnosis of HIV infection
* Active chronic hepatitis B or C infection
* Subjects who have clinically significant abnormality/finding from examination, tests, or history that may compromise subject safety, specifically any history of cardiac, renal or hepatic impairment
* Subjects with an abnormal ECG
* Persistent arterial hypotension, with average SBP readings of ≤95 mmHg
* Persistent elevation of blood pressure, with average SBP readings of ≥160 mmHg or average DBP readings of ≥100 mmHg
* Pregnant or lactating females
* Participation in another clinical study in 28 days prior to Screening Visit
* Evidence of clinically significant renal, hepatic, cardiac, pulmonary (apart from asthma) or metabolic dysfunction, e.g. diabetes mellitus, thyrotoxicosis, uncorrectable hypokalaemia, or predisposition to low levels of serum potassium
* Current/history of drug/alcohol abuse/dependence per WHO criteria
* Inability to communicate well w/investigator
* Donation of ≥450 mL of blood/blood products within previous 3 months prior to screening
* History of allergy/intolerance/contraindications to corticosteroids/lactose, or severe allergy to milk proteins
* Consumption of alcohol- or caffeine-containing foods/beverages from midnight before or during Screening Visit
* History of medically diagnosed chronic respiratory diseases other than asthma (e.g. chronic obstructive pulmonary disease, ABPA in the absence of asthma)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (11):
  - Vectura Clinical Trial Site 01001, Los Angeles, California
  - Vectura Clinial Trial Site 01005, Denver, Colorado
  - Vectura Clinical Trial Site 01006, Celebration, Florida
  - Vectura Clinical Trial Site 01015, Hialeah, Florida
  - Vectura Clinical Trial Site 01012, Miami Lakes, Florida
  - Vectura Clinical Trial Site 01014, Orlando, Florida
  - Vectura Clinical Trial Site 01003, Tampa, Florida
  - Vectura Clinical Trial Site 01011, St Louis, Missouri
  - Vectura Clinical Trial Site 01013, Jersey City, New Jersey
  - Vectura Clinical Trial Site 01004, The Bronx, New York
  - Vectura Clinical Trial Site 01007, El Paso, Texas
- Bulgaria (8):
  - Vectura Clinical Trial Site 08006, Rousse
  - Vectura Clinical Trial Site 08005, Sofia
  - Vectura Clinical Trial Site 08001, Sofia
  - Vectura Clinical Trial Site 08003, Sofia
  - Vectura Clinical Trial Site 08007, Sofia
  - Vectura Clinical Trial Site 08004, Sofia
  - Vectura Clinical Trial Site 08002, Stara Zagora
  - Vectura Clinical Trial Site 08008, Varna
- Germany (9):
  - Vectura Clinical Trial Site 03006, Berlin
  - Vectura Clinical Trial Site 03009, Berlin
  - Vectura Clinical Trial Site 03004, Bonn
  - Vectura Clinical Trial Site 03008, Donaustauf
  - Vectura Clinical Trial Site 03003, Dortmund
  - Vectura Clinical Trial Site 03007, Geesthacht
  - Vectura Clinical Trial Site 03001, Hamburg
  - Vectura Clinical Trial Site 03005, Heidelberg
  - Vectura Clinical Trial Site 03002, Rüdersdorf
- Hungary (5):
  - Vectura Clinical Trial Site 04001, Budapest
  - Vectura Clinical Trial Site 04004, Budapest
  - Vectura Clinical Trial Site 04003, Debrecen
  - Vectura Clinical Trial Site 04002, Rakoczi
  - Vectura Clinical Trial Site 04005, Rakoczi
- Poland (11):
  - Vectura Clinical Trial Site 05008, Bialystok
  - Vectura Clinical Trial Site 05002, Bialystok
  - Vectura Clinical Trial Site 05010, Bialystok
  - Vectura Clinical Trial Site 05011, Krakow
  - Vectura Clinical Trial Site 05001, Lodz
  - Vectura Clinical Trial Site 05006, Lodz
  - Vectura Clinical Trial Site 05005, Lublin
  - Vectura Clinical Trial Site 05007, Tarnów
  - Vectura Clinical Trial Site 05003, Warsaw
  - Vectura Clinical Trial Site 05009, Wroclaw
  - Vectura Clinical Trial Site 05004, Zawadzkie
- Romania (14):
  - Vectura Clinical Trial Site 07001, Brasov
  - Vectura Clinical Trial Site 07008, Bucharest
  - Vectura Clinical Trial Site 07005, Bucharest
  - Vectura Clinical Trial Site 07013, Bucharest
  - Vectura Clinical Trial Site 07003, Bucharest
  - Vectura Clinical Trial Site 07006, Cluj-Napoca
  - Vectura Clinical Trial Site 07007, Cluj-Napoca
  - Vectura Clinical Trial Site 07009, Cluj-Napoca
  - Vectura Clinical Trial Site 07014, Craiova
  - Vectura Clinical Trial Site 07002, Iași
  - Vectura Clinical Trial Site 07004, Marghita
  - Vectura Clinical Trial Site 07010, Sadu
  - Vectura Clinical Trial Site 07012, Târgu Mureş
  - Vectura Clinicl Trial Site 07011, Timuș
- Ukraine (14):
  - Vectura Clinical Trial Site 06013, AR Crimea
  - Vectura Clinical Trial Site 06009, Donetsk
  - Vectura Clinical Trial Site 06012, Ivano-Frankivsk
  - Vectura Clinical Trial Site 06010, Kharkiv
  - Vectura Clinical Trial Site 06001, Kharkiv
  - Vectura Clinical Trial Site 06004, Kharkiv
  - Vectura Clinical Trial Site 06006, Kyiv
  - Vectura Clinical Trial Site 06002, Kyiv
  - Vectura Clinical Trial Site 06015, Kyiv
  - Vectura Clinical Trial Site 06003, Kyviv
  - Vectura Clinical Trial Site 06008, Mykolaiv
  - Vectura Clinical Trial Site 06011, Vinnitsa
  - Vectura Clinical Trial Site 06007, Zaporizhzhia
  - Vectura Clinical Trial Site 06014, Zaporizhzhya
- United Kingdom (5):
  - Vectura Clinical Trial Site 02003, Cottingham, Hull
  - Vectura Clinical Trial site 02002, Birmingham
  - Vectura Clinical Trial Site 02004, Manchester
  - Vectura Clinical Trial Site 02001, Newcastle
  - Vectura Clinical Trial Site 02005, Nottingham

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 197 subjects were randomised and 196 received at least one dose of study drug; 1 subject was randomised but not treated.
Groups:
- Dose 1 VR506 50 mcg; Dose 2 VR506 250 mcg; Dose 3 VR506 500 mcg: VR506 inhalation powder delivered via a new dry powder inhaler device
  VR506: VR506 inhalation powder delivered via a new dry powder inhaler device
Period: Overall Study
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
Started | 62 | 71 | 63
Full Anaylsis Set | 62 | 71 | 63
Completed | 57 | 56 | 48
Not Completed | 5 | 15 | 15
Not completed — Could not use e-diary correctly | 0 | 1 | 1
Not completed — Randomised without baseline values | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 4 | 0
Not completed — Treatment period withdrawal criteria met | 4 | 8 | 9
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — OCS bursts occured, discontinued in line | 1 | 0 | 0
Not completed — Non-compliance on using e-diary | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg | Total
Number analyzed (Participants) | 62 | 71 | 63 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 62 | 70 | 63 | 195
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 45 | 42 | 127
  Male | 22 | 26 | 21 | 69
Region of Enrollment [Number; unit: participants]
  Romania | 16 | 17 | 16 | 49
  Hungary | 3 | 3 | 4 | 10
  United States | 2 | 4 | 4 | 10
  Ukraine | 15 | 18 | 14 | 47
  Poland | 15 | 18 | 16 | 49
  United Kingdom | 1 | 1 | 0 | 2
  Bulgaria | 6 | 7 | 6 | 19
  Germany | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Prednisone/Prednisolone Dose for Analysis (PDA) at End of Study (Week 16)
Description: The mean asthma control prednisone/prednisolone dose at end of study (week 16)
Time Frame: 16 weeks
Population: The Full Analysis Set (FAS) was analyzed, however 7 subjects are not included because they had no OCS dose adjustment assessment post-randomisation, and baseline values were not carried forward.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
Number analyzed (Participants) | 61 | 70 | 58
mg | 4.55 (6.85) | 4.31 (7.38) | 3.97 (6.21)
Statistical Analysis 1: Comparison: Dose 1 VR506 50 mcg vs Dose 2 VR506 250 mcg vs Dose 3 VR506 500 mcg; Test type: Superiority; p = 0.772, ANCOVA

2. Secondary Outcome: Mean Change From Start of Treatment Baseline to End of Study (Week 16) for In-clinic Morning Pre-Dose Forced Expiratory Volume In 1 Second (FEV1)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
Number analyzed (Participants) | 62 | 71 | 63
Liters | 0.06 (0.4) | 0.02 (0.31) | 0.06 (0.35)
Statistical Analysis 1: Comparison: Dose 1 VR506 50 mcg vs Dose 2 VR506 250 mcg vs Dose 3 VR506 500 mcg; Test type: Superiority; p = 0.891, ANCOVA

3. Secondary Outcome: Mean Change From Start of Treatment Baseline to End of Study (Week 16) for Asthma Control Questionnaire (ACQ-5) Mean Total Score
Description: Change from baseline to end of study (week 16) in 5 item asthma control questionnaire (ACQ-5) mean total score (range 0 (better) to 6 (worse)). The mean total score is calculated as the mean for each subject at each visit of 5 questions, each scored from 0 (better) to 6 (worse).
Time Frame: Baseline and 16 weeks
Population: Full Analysis Set was analyzed, but number of patients represents subjects with both start of treatment baseline value and end of treatment value where a Last Observation Carried Forward (LOCF) approach was used to impute values of missing post-baseline visits; 1 subject had no post-dose ACQ-5 assessment, baseline value was not carried forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
Number analyzed (Participants) | 62 | 70 | 63
score on a scale | -0.67 (0.98) | -0.77 (1.15) | -0.39 (0.89)
Statistical Analysis 1: Comparison: Dose 1 VR506 50 mcg vs Dose 2 VR506 250 mcg vs Dose 3 VR506 500 mcg; Test type: Superiority; p = 0.066, ANCOVA

4. Secondary Outcome: Mean Change From Start of Treatment Baseline to End of Study (Week 16) for In-clinic Weekly Morning Pre-dose Peak Expiratory Flow (PEF)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
Number analyzed (Participants) | 62 | 71 | 63
L/min | 2 (45.7) | 20.1 (51.7) | 6.1 (53.5)
Statistical Analysis 1: Comparison: Dose 1 VR506 50 mcg vs Dose 2 VR506 250 mcg vs Dose 3 VR506 500 mcg; Test type: Superiority; p = 0.063, ANCOVA

5. Secondary Outcome: Mean Change From Start of Treatment Baseline to End of Study (Week 16) for Weekly Average Asthma Night-time Symptom Score
Description: To measure the change from baseline to end of study for the weekly mean asthma night time symptom score, scored from 0 (not at all bothered) to 6 (severely bothered).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
Number analyzed (Participants) | 62 | 71 | 63
score on a scale | -0.3 (1) | -0.6 (1) | -0.2 (1)
Statistical Analysis 1: Comparison: Dose 1 VR506 50 mcg vs Dose 2 VR506 250 mcg vs Dose 3 VR506 500 mcg; Test type: Superiority; p = 0.054, ANCOVA

6. Secondary Outcome: Number of Participants With Withdrawals Due to Worsening of Asthma
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
Number analyzed (Participants) | 62 | 71 | 63
Participants | 4 | 11 | 8
Statistical Analysis 1: Comparison: Dose 1 VR506 50 mcg vs Dose 2 VR506 250 mcg; Test type: Superiority; p = 0.168, Fisher Exact
Statistical Analysis 2: Comparison: Dose 1 VR506 50 mcg vs Dose 3 VR506 500 mcg; Test type: Superiority; p = 0.363, Fisher Exact
Statistical Analysis 3: Comparison: Dose 2 VR506 250 mcg vs Dose 3 VR506 500 mcg; Test type: Superiority; p = 0.805, Fisher Exact

7. Secondary Outcome: Assessment of Acceptability of the Device
Description: Percentage of subjects that overall found it very easy or fairly easy to use the inhaler, based on inhaler acceptability questionnaire
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
Number analyzed (Participants) | 62 | 71 | 63
Participants
  Very easy | 40 | 49 | 38
  Fairly easy | 21 | 21 | 21
  Missing | 1 | 1 | 4

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Dose 1 VR506 50 mcg | Dose 2 VR506 250 mcg | Dose 3 VR506 500 mcg
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/71 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/71 | 0/63
Other Adverse Events (participants affected / at risk) | 21/62 | 33/71 | 25/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 VR506 50 mcg (N=62) | Dose 2 VR506 250 mcg (N=71) | Dose 3 VR506 500 mcg (N=63)
Asthma (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 26 (35) | 12 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 2 (3)
Acute sinusitis (Infections and infestations) | 0 (0) | 3 (4) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Phyaryngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystisis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngitis Fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis Streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Aspartate Aminotransferase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Middle Ear Effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Vectura's agreements with its investigators may vary. Publication may be delayed for Sponsor review and revisions/deletions can be required. Furthermore, a delay to publication may be required by the Sponsor in order to take steps to protect its proprietary information and/or intellectual property rights.